CLINICAL TRIAL: NCT06692374
Title: Smartwatch-based Automated Cardiac Arrest Detection and Activation of the Emergency Medical Chain: Validation in a Home Setting
Brief Title: Automated Cardiac Arrest Detection and Alerting in Daily Life
Acronym: DETECT-4b
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Corsano Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: 116424
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Arrest (CA); Sudden Death, Cardiac
Keywords: Automated cardiac arrest detection; Wearable; Photoplethysmography; Sudden Cardiac Death
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Surviving a cardiac arrest that happens outside the hospital depends on quickly recognizing the event and immediately starting CPR. Survival rates have improved when cardiac arrest is witnessed, but when it isn't, help often arrives too late. Wearable biosensors, like special wristbands, could detect cardiac arrest automatically and alert emergency responders, providing faster help.

In the already finished DETECT-1 study, the investigators developed a system that uses wrist-worn sensors to identify cardiac arrest. The goal of the current study is to test how well this system works in people who have an implantable cardioverter defibrillator (ICD). An ICD is a device that monitors and treats dangerous heart rhythms. Study participants will wear a medical wristband with sensors that monitor the heartrate and movement during their daily activities to see if the system accurately detects cardiac arrest.

DETAILED DESCRIPTION:
Survival from out-of-hospital cardiac arrest (OHCA) depends on fast recognition of cardiac arrest and immediate initiation of cardiopulmonary resuscitation (CPR). While survival chances for witnessed OHCA have increased, unwitnessed cases still often receive help too late. Wearable biosensor technology with the functionality of automated cardiac arrest detection and activation of the emergency medical chain would offer a potential solution to provide early help. In the recently published DETECT-1 study, an algorithm for automated cardiac arrest detection using wrist-derived photoplethysmography (PPG) was recently developed.

The current study is a prospective multicenter observational cohort study to validate the sensitivity of the developed cardiac arrest detection algorithm in patients with an implantable cardioverter defibrillator (ICD) during daily life. The study population includes patients with an ICD. Study participants will wear a medical wristband with PPG and accelerometer sensors during daily life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implantable cardioverter defibrillator (ICD)
* Age 18 years or older
* Fitting the wristband
* In possession of a smartphone that is compatible with the wristband

Exclusion Criteria:

* Known hemodynamically relevant bilateral subclavian artery stenosis
* Medical issues that interfere with wearing of the wristband (e.g. skin disorders)
* Insufficient skills to operate with the device/app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with an ICD.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for cardiac arrest detection | From the time of enrollment to the end of the wearing period of the wristband (maximal two years)
  The number of correctly identified cardiac arrest events by the algorithm devided by the total number of cardiac arrest events.

SECONDARY OUTCOMES:
Positive predictive value for cardiac arrest detection | From the time of enrollment to the end of the wearing period of the wristband (maximal two years)
  The number of true positives devided by the sum of the true positives and false positive cardiac arrest alarms
False positive alarm rate | From the time of enrollment to the end of the wearing period of the wristband (maximal two years)
  Expressed as the number of false positive non-cancelled cardiac arrest alarms per user year

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Pseudomynized data from the wristband will be made available on a data repository under restricted access.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be made available when results of the study are published, for 15 years.

REFERENCES:
- [Result] Edgar R, Scholte NTB, Ebrahimkheil K, Brouwer MA, Beukema RJ, Mafi-Rad M, Vernooy K, Yap SC, Ronner E, van Mieghem N, Boersma E, Stas PC, van Royen N, Bonnes JL. Automated cardiac arrest detection using a photoplethysmography wristband: algorithm development and validation in patients with induced circulatory arrest in the DETECT-1 study. Lancet Digit Health. 2024 Mar;6(3):e201-e210. doi: 10.1016/S2589-7500(23)00249-2. PMID 38395540
- See also: Related Info — https://detect-study.com/en/